CLINICAL TRIAL: NCT03489499
Title: Genetic Variants and Postoperative Pain
Status: Recruiting | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 041/09c Schmerz
Record Dates: First submitted 2018-03-29; First posted 2018-04-05 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Pain; Analgesia; Surgical Procedure, Operative
Keywords: postoperative pain; analgesics; patient reported outcome; pain related impairment; genetic association study
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood (plasma and cells) or mucosal swab
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- All patients: Patients undergoing elective surgery with anesthesia

SUMMARY:
Prospective observational study to analyse patients' pain related outcome after surgery and ist association to genetic variants and non-genetic variables.

DETAILED DESCRIPTION:
Background

Severe acute pain as well as long-lasting pain after surgery and pain-related interference of daily activities are frequent. Some risk factors for severe pain after surgery in adults have been described, e.g. younger age and pre-existing chronic pain. The question arises whether a specific genetic background is related to an unfavorable pain outcome.

Objective

The aim of this study is to investigate clinical and genetic variables and their possible association to severe acute postoperative pain, higher analgesic consumption and the development of chronic postsurgical pain.

Methods

Prospective observational study investigating clinical, patient related, surgery related and anesthesia related variables as well as genetic variants and their possible association to patients' pain related outcome after surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Written informed consent
* Elective surgery
* Patients' ability to understand the purpose of the study

Exclusion Criteria

* No informed consent
* Cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients scheduled for elective surgery
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2011-01-02 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Pain related impairment after surgery and its association to genetic and non-genetic variables | day of surgery up to 1 year after surgery
  Measured by the International Pain Outcomes Questionnaire, the Brief Pain Inventory (BPI): Numeric rating scale for pain intensities, affective and physical interference; Composite score = pain interference total scores (PITS scale 0-10) resulting in no interference (PITS=0), mild interference (PITS >0 and <2), moderate interference (PITS 2-5) and severe interference (PITS >5)

SECONDARY OUTCOMES:
Association of genetic and non-genetic variables with analgesic consumption | day of surgery up to one year after surgery
  analgesic consumption
Association of genetic and non-genetic variables with pain related outcome of patients 1 year after surgery | Up to one year after surgery
  Measured by the Brief Pain Inventory (BPI) as pain interference total score PITS scale 0-10) resulting in no interference (PITS=0), mild interference (PITS >0 and <2), moderate interference (PITS 2-5) and severe interference (PITS >5).
  Change of pain related impairment over time (before surgery, 2 days after surgery, 6 and 12 months after surgery)
Association of genetic and non-genetic variables with chronic neuropathic postsurgical pain | up to one year after surgery
  Measured by a neuropathic pain questionnaire (number of neuropathic symptoms; at least three neuropathic symptoms are categorized as positive)

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Stamer, Prof. MD, Study Chair — Department of Anaestheisolpogy + Pain Medicine, Inselspital, University of Bern; Ulrike M Stamer, MD, Principal Investigator — Department of Anaesthesiology and Pain Medicine, Inselspital, University of Bern
Locations (1):
- Department of Anaesthesiology and Pain Medicine, Inselspital, University of Bern, Bern, Switzerland